CLINICAL TRIAL: NCT06579300
Title: A Phase 1 Multiple Ascending Dose, Drug-Drug Interaction, and Asian Pharmacokinetic Study of ABBV-1088
Brief Title: A Study to Assess Multiple Ascending Dose, Drug-Drug Interaction, and Asian Pharmacokinetic Study of ABBV-1088
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: M24-931
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; ABBV-1088; Itraconazole
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (14):
- Part 1: Group 1 ABBV-1088 Dose A (Experimental): Participants will receive ABBV-1088 dose A for 7 days
  Interventions: Drug: ABBV-1088
- Part 1: Group 1 Placebo (Experimental): Participants will receive placebo for 7 days
  Interventions: Drug: Placebo for ABBV-1088
- Part 1: Group 2 ABBV-1088 Dose B (Experimental): Participants will receive ABBV-1088 dose B for 21 days
  Interventions: Drug: ABBV-1088
- Part 1: Group 2 Placebo (Experimental): Participants will receive placebo for 21 days
  Interventions: Drug: Placebo for ABBV-1088
- Part 1: Group 3 ABBV-1088 Dose C (Experimental): Participants will receive ABBV-1088 dose C for 7 days
  Interventions: Drug: ABBV-1088
- Part 1: Group 3 Placebo (Experimental): Participants will receive placebo for 7 days
  Interventions: Drug: Placebo for ABBV-1088
- Part 1: Group 4 ABBV-1088 Dose D (Experimental): Participants will receive ABBV-1088 dose D for 21 days
  Interventions: Drug: ABBV-1088
- Part 1: Group 4 Placebo (Experimental): Participants will receive placebo for 21 days
  Interventions: Drug: Placebo for ABBV-1088
- Part 1: Group 5 ABBV-1088 Dose D (Experimental): Participants older than 60 years of age will receive ABBV-1088 dose D for 21 days
  Interventions: Drug: ABBV-1088
- Part 1: Group 5 Placebo (Experimental): Participants older than 60 years of age will receive placebo for 21 days
  Interventions: Drug: Placebo for ABBV-1088
- Part 2: Period 1 ABBV-1088 Dose A (Experimental): Participants will receive ABBV-1088 Dose A on day 1
  Interventions: Drug: ABBV-1088
- Part 2: Period 2 ABBV-1088 Dose A with ITZ (Experimental): Participants will receive ABBV-1088 dose A on day 4 with itraconazole (ITZ) for 10 days
  Interventions: Drug: ABBV-1088; Drug: Itraconazole (ITZ)
- Part 3: Group 1 ABBV-1088 Han Chinese Participants (Experimental): Han Chinese participants will receive ABBV-1088 dose E on day 1
  Interventions: Drug: ABBV-1088
- Part 3: Group 2 ABBV-1088 Japanese Participants (Experimental): Japanese participants will receive ABBV-1088 dose E on day 1
  Interventions: Drug: ABBV-1088

INTERVENTIONS:
Drug: ABBV-1088 — Oral Capsule
  Arms: Part 1: Group 1 ABBV-1088 Dose A; Part 1: Group 2 ABBV-1088 Dose B; Part 1: Group 3 ABBV-1088 Dose C; Part 1: Group 4 ABBV-1088 Dose D; Part 1: Group 5 ABBV-1088 Dose D; Part 2: Period 1 ABBV-1088 Dose A; Part 2: Period 2 ABBV-1088 Dose A with ITZ; Part 3: Group 1 ABBV-1088 Han Chinese Participants; Part 3: Group 2 ABBV-1088 Japanese Participants
Drug: Placebo for ABBV-1088 — Oral Capsule
  Arms: Part 1: Group 1 Placebo; Part 1: Group 2 Placebo; Part 1: Group 3 Placebo; Part 1: Group 4 Placebo; Part 1: Group 5 Placebo
Drug: Itraconazole (ITZ) — Oral Capsule
  Arms: Part 2: Period 2 ABBV-1088 Dose A with ITZ

SUMMARY:
This study will assess the safety, tolerability, and pharmacokinetics of ABBV-1088 in healthy adult Western, Han-Chinese and Japanese participants. This study will also assess drug-drug interaction between itraconazole and ABBV-1088 in healthy adult Western participants.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) is > = 18.0 to < = 32.0 kg/m^2 after rounded to the tenths decimal, at Screening and upon confinement.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG.
* Part 3 Only: Han Chinese Participant must be first-or second-generation Han Chinese of full Chinese parentage. First-generation participants will have been born in China to two participants and four grandparents also born in China of full Chinese descent. Second-generation participants born outside of China must have two parents and four grandparents born in China of full Chinese descent. Participants must maintain a typical Chinese lifestyle, including consuming a typical Chinese diet. OR
* Japanese Participant must be first-or second-generation Japanese of full Japanese parentage. First-generation participants will have been born in Japan to two parents and four grandparents also born in Japan of full Japanese descent. Second-generation participants born outside of Japan must have two parents and four grandparents born in Japan of full Japanese descent. All participants must maintain a typical Japanese lifestyle, including consuming a typical Japanese diet.

Exclusion Criteria:

* Part 1 (Groups 1-4), Part 2 and Part 3: History of any clinically significant neurological, respiratory (except mild asthma as a child), endocrine, metabolic, renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.
* History of suicidal ideation within one year prior to study drug administration as evidenced by answering "yes" to questions 4 or 5 on the suicidal ideation portion of the Columbia Suicide Severity Rating Scale (C-SSRS) completed at Screening, or any history of suicide attempts within the last two years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Part 1, 2 and 3: Maximum Plasma Concentration (Cmax) of ABBV-1088 | Up to approximately 24 days
  Cmax of ABBV-1088
Part 1, 2 and 3: Time to Cmax (Tmax) of ABBV-1088 | Up to approximately 24 days
  Tmax of ABBV-1088
Part 1, 2 and 3: Terminal Phase Elimination Rate Constant (Beta) of ABBV-1088 | Up to approximately 24 days
  Terminal phase elimination rate constant (beta) of ABBV-1088
Part 1, 2 and 3: Terminal Phase Elimination Half-Life (t1/2) of ABBV-1088 | Up to approximately 24 days
  Terminal phase elimination half-life of ABBV-1088
Part 2 and 3: Area Under the Concentration-Time Curve from Time 0 to Time t (AUCt) of ABBV-1088 | Up to approximately 24 days
  AUCt of ABBV-1088
Part 2 and 3: Area Under the Concentration-Time Curve from Time 0 to Infinity (AUCinf) of ABBV-1088 | Up to approximately 24 days
  AUCinf of ABBV-1088
Number of Participants with Adverse Events (AEs) | Up to approximately 54 days
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study
Part 1: Trough Concentration (Ctrough) of ABBV-1088 | Up to approximately 24 days
  Ctrough of of ABBV-1088
Part 1: Area Under the Plasma Concentration-time Curve (AUC) for the First and Final Dose Intervals (AUCtau) | Up to approximately 24 days
  The area under the plasma concentration-time curve over a dosing interval of tau (AUCtau).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (2):
- United States (2):
  - CenExel ACT- Anaheim Clinical Trials /ID# 276423, Anaheim, California
  - Acpru /Id# 270552, Grayslake, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-931